CLINICAL TRIAL: NCT05754723
Title: Developing, Administering, and Evaluating Online Psychotherapy and Psychoeducation Programs for Postsecondary Students Within a Regional Mental Health Hub in Ontario, Canada Using AI-assisted Online Interventions
Brief Title: Using an Online Psychotherapy Program and AI-assisted Interventions for Postsecondary Student Mental Health
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was not obtained
Sponsor: Dr. Nazanin Alavi (Other)
Responsible Party: Sponsor-Investigator, Dr. Nazanin Alavi, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6034514
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Mental Health Issue
Keywords: Student; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Aim 1 will assess post-secondary students' current mental health needs, through surveys and focus groups. Aims 2 and 3 will use the findings from the surveys and focus groups to inform the development of 6-week psychoeducation and 12-week diagnosis-specific e-CBT programs. The psychoeducation program will be followed by 6-months of AI-assisted journaling exercises to monitor the student's mental health and determine whether they would benefit from stepping up their care to receive the diagnosis-specific e-CBT program. Aims 4 and 5 will determine the efficacy and cost-effectiveness of the online psychoeducation and diagnosis-specific e-CBT programs by comparing them to treatment as usual. Aims 6 and 7 will use the data to monitor the success and fidelity of the programs using surveys and focus groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-Psychotherapy (Experimental): Participants in the treatment group will receive access to the hub's services which begin with six weeks of online psychoeducation. Participants will be recruited through on-campus flyers, advertisements and wellness-center announcements, media advertisements, expert end-user referrals, and self-referrals. Participants will be excluded if they have active psychosis, acute mania, and/or active suicidal or homicidal ideation, and have received psychoeducation or psychotherapy like that offered by our proposed hub in the past six months. Participants with high disorder severity will be referred to other community resources determined by clinicians and therapists on the research team.
  Interventions: Behavioral: e-Psychotherapy/Psychoeducation
- Treatment as Usual (No Intervention): TAU will consist of medications, regular physician or clinician visits, referrals or consultations that are conducted outside of the current research study.

INTERVENTIONS:
Behavioral: e-Psychotherapy/Psychoeducation — Participants will receive six weekly self-guided psychoeducation sessions. Then, after 6 weeks participants will complete monthly clinical questionnaires for 6 months. Also, participants will begin bi-weekly journaling exercises for 6 months. Based on the journaling entries, if the AI algorithm detects MDD, GAD, SAD or ADHD that requires treatment will make a referral to the diagnosis-specific e-CBT (MDD, GAD, SAD or ADHD). If after 6 months, no referral decision is made by the AI algorithm no extra follow-up will be provided. Once the AI makes a referral recommendation, participants will be placed in a diagnosis-specific e-CBT program specific to the diagnosis determined by the AI algorithm (MDD, GAD, SAD, or ADHD). The asynchronous e-CBT programs will consist of 12 weekly modules and homework. Weekly homework is reviewed by a therapist, who will provide personalized feedback based on the participant's preferred method (i.e., text, video, or audio).
  Arms: e-Psychotherapy

SUMMARY:
The prevalence of mental health challenges and disorders in post-secondary students, demands accessible and efficacious care. Online psychotherapy and psychoeducation programs have shown significant effectiveness in mitigating the risk and clinical symptoms of various mental health disorders. Additionally, artificial intelligence (AI) has become an accessible, effective, and scalable tool supporting the delivery of healthcare. Therefore, the primary objective of this study is to develop an AI-driven online mental health care hub in the Kingston, Frontenac, Lennox & Addington region for post-secondary students. . This hub will deliver equitable, efficacious, and cost-effective online psychoeducation and psychotherapy in the form of online diagnosis-specific cognitive behavioural therapy (e-CBT). The hub's virtual design aims to adequately address existing gaps in the mental healthcare of these individuals and alleviate the burden placed on mental health services in Canada. Using a rigorous implementation framework, the development of this hub is designed as a multiphase study with three phases. (1) Pre-adoption phase: will assess post-secondary students' current mental health landscape through surveys and focus groups. This information will be used in the development of our online psychoeducation and diagnosis-specific e-CBT programs. (2) Delivery phase: will determine the efficacy and cost-effectiveness of the online psychoeducation and diagnosis-specific e-CBT programs by comparing them to treatment as usual. (3) Post-adoption phase: the collected data from these programs will be analyzed and shared with key stakeholders to guide continuous program scaling and improvement.

DETAILED DESCRIPTION:
The proposed regional mental healthcare hub aims to deliver equitable, efficacious, and cost-effective AI-driven online psychoeducation and diagnosis-specific online cognitive behavioural therapy (e-CBT) programs for post-secondary students in the Kingston, Frontenac, Lennox & Addington (KFL&A) region. The initiative will target a broad population of students ranging from those interested in learning more about mental health (online psychoeducation program) to those seeking additional help for their psychiatric symptoms (e-CBT program). Our research team is strongly experienced in designing effective AI-assisted online psychoeducation and diagnosis-specific e-CBT programs for various mental health conditions in diverse populations. Therefore, being as effective as in-person methods of healthcare delivery, it is hypothesized that our online interventions disseminated via a robust implementation science and community collaboration strategy will be a feasible, cost-effective, and pragmatic solution to address accessibility issues with post-secondary student mental healthcare.

The proposed mental health hub will offer a comprehensive care model using a stepped-care approach. Its implementation will be guided by a rigorous approach involving seven aims divided into three phases (pre-adoption, delivery, and post-adoption phases). (1) Pre-adoption phase: will assess post-secondary students' current mental health landscape through surveys and focus groups (Aim 1). This information will be used in the development of a 6-week online psychoeducation (Aim 2) and 12-week diagnosis-specific e-CBT (Aim 3) programs. The psychoeducation program will be followed by 6-months of AI-assisted journaling exercises to monitor the student's mental health and determine whether they would benefit from stepping up their care to receive the diagnosis-specific e-CBT program. The diagnosis-specific e-CBT programs will be adapted from prior clinically validated and diagnosis-specific psychotherapy modules developed by the lab. Four diagnosis-specific modules will support the most common mental health disorders in students (GAD, SAD, MDD and ADHD), as indicated by previous studies and the research team's cross-sectional survey of students in Ontario, Canada. Both programs will be delivered through the Online Psychotherapy Tool (OPTT) - a secure cloud-based platform co-developed by the PI that offers online mental health interventions. (2) Delivery phase: will determine the efficacy and cost-effectiveness of the online psychoeducation (Aim 4) and diagnosis-specific e-CBT (Aim 5) programs by comparing them to treatment, as usual, using validated clinical assessment tools. (3) Post-adoption phase: will use the collected data to monitor the success and fidelity of the programs using surveys and focus groups (Aim 6), and to build capacity and scale the project to other Canadian municipalities (Aim 7). As such, in contrast to other initiatives that target student mental health, this will be the first to involve students and end-users in all phases, from conception to implementation.

The digital nature of this healthcare program and the implementation of AI technology results in new solutions that enable easier accessibility and broader reach to individuals in significant need of mental healthcare services. Therefore, to support the development of these mental healthcare resources, the research team has assembled a diverse, cross-functional interdisciplinary team of community leaders, including researchers, clinicians, health decision-makers, and end-users. Ultimately, leveraging the extensive expertise of a cross-functional research team, the objective of the study is to develop and implement a successful and effective digital care plan with the potential to improve post-secondary student mental health care substantially.

ELIGIBILITY:
Inclusion Criteria:

* post-secondary students enrolled in institutions of interest
* the ability to provide informed consent
* the ability to speak and read English
* consistent and reliable access to the internet

Exclusion Criteria:

- N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Change in anxiety severity (GAD-7) | weeks 0, 3, 6, follow-up 1, 2, 3, 4, 5, 6 months
  Generalized anxiety disorder - 7 item (GAD-7) questionnaire. Increase in score dictates increase in severity. Scale of 0-3
Change in depression severity (PHQ-9) | weeks 0, 3, 6, follow-up 1, 2, 3, 4, 5, 6 months
  Patient Health Questionnaire - 9 item (PHQ-9). Increase in score dictates increase in severity. Scale of 0-3 on each question.
Change in depression severity (QIDS) | weeks 0, 3, 6, follow-up 1, 2, 3, 4, 5, 6 months
  Quick Inventory of Depressive Symptomatology (QIDS). Increase in score dictates increase in severity. Scale of 0-3 on each question
Change in stress severity (DASS-42) | weeks 0, 3, 6, follow-up 1, 2, 3, 4, 5, 6 months
  Depression Anxiety Stress Scale-42 (DASS-42). Increase in score dictates increase in severity. Scale of 0-3 on each question.
Change in quality of life (AQoL-8D) | weeks 0, 3, 6, follow-up 1, 2, 3, 4, 5, 6 months
  Assessment of Quality of Life-8D (AQoL-8D). Increase in score dictates increase in quality of life (improvement). Scale of 0-5 on each question.
Change in resilience (RS-14) | weeks 0, 3, 6, follow-up 1, 2, 3, 4, 5, 6 months
  Resilience Scale-14 (RS-14). Increase in score dictates increase in resilience (improvement). Scale of 0-7 on each question
Change in social anxiety severity (LSAS) | weeks 0, 3, 6, follow-up 1, 2, 3, 4, 5, 6 months
  Liebowitz Social Anxiety Scale (LSAS). Increase in score dictates increase in anxiety severity. Scale of 0-3 on each question.
Change in ADHD severity (ASRS) | weeks 0, 3, 6, follow-up 1, 2, 3, 4, 5, 6 months
  Adult ADHD Self-Report Scale (ASRS). Increase in score dictates increase in ADHD symptom severity. Scale of 0-5 on each question.

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Alavi, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request
Supporting Information: Study Protocol
Time Frame: Post-study
Access Criteria: Available upon request to researchers